CLINICAL TRIAL: NCT05956938
Title: Effect of Training Using Action Video Games and Stroboscopic Glasses on Dynamic Visual Acuity.
Brief Title: Effect of Action Video Games and Stroboscopic Glasses on Dynamic Visual Acuity.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Politècnica de Catalunya (Other)
Responsible Party: Principal Investigator, Marc Argilés Sans, Principal Investigator, Universitat Politècnica de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAD1
Record Dates: First submitted 2023-07-05; First posted 2023-07-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Visual Acuity
Keywords: Dynamic visual acuity; Action video games; Stroboscopic glasses

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Action Video game Group (Experimental): A one-hour training session will be held, divided into 2 30-minute sessions over 2 days. Each session will take into account an increase in the difficulty of the task gradually based on the nature of the video game. The video game selected will be ContraIII: Alien Wars, from the Nintendo Mini Classic console.
  Interventions: Device: Action Video Game
- Stroboscopic Glasses Group (Experimental): A one-hour training session will be held, divided into 2 30-minute sessions over 2 days. Each session will take into account a gradual increase in the difficulty of the task, divided into three visuomotor and anticipation components (ball size, type of trajectory and distance from the stimulus). The training sessions will consist of 2 series, and will be based on passing a ball between two people. Every 60 passes the flicker level of the glasses will increase, starting with level 1 (6hz) and ending at level 6 (1.75hz).
  Interventions: Device: Stroboscopic Glasses
- Control Group (No Intervention): Participants in the control group will watch 1 video clip/series/film of 1 hour duration on a television located at least 1.5 meters away.

INTERVENTIONS:
Device: Stroboscopic Glasses — A one-hour training session will be held, divided into 2 30-minute sessions over 2 days. Each session will take into account a gradual increase in the difficulty of the task, divided into three visuomotor and anticipation components (ball size, type of trajectory and distance from the stimulus).
  The training sessions will consist of 2 series, and will be based on passing a ball between two people. Every 60 passes the flicker level of the glasses will increase, starting with level 1 (6hz) and ending at level 6 (1.75hz)
  Arms: Stroboscopic Glasses Group
Device: Action Video Game — A one-hour training session will be held, divided into 2 30-minute sessions over 2 days. Each session will take into account an increase in the difficulty of the task gradually based on the nature of the video game. The video game selected will be ContraIII: Alien Wars, from the Nintendo Mini Classic console.
  Arms: Action Video game Group

SUMMARY:
The study aims to observe the possible improvement of performance in dynamic visual acuity (DVA), in terms of speed and trajectory, comparing training using action video games and strobe glasses. The results will allow us to understand which visual training is more beneficial for improving dynamic visual acuity in athletes.

DETAILED DESCRIPTION:
During the last years there have been several investigations related to the effect of action video games (VA) on the visual system, specifically perceptual and cognitive processes. These investigations indicate that playing VA can be a powerful tool for improving visuo-spatial attention, visuo-motor control, and reaction time. On the other hand, certain studies indicate that the use of stroboscopic glasses can help improve sports performance, and especially dynamic visual acuity , as well as various visual performance skills. The study aims to observe the possible improvement of performance in dynamic visual acuity (DVA), in terms of speed and trajectory, comparing training using action video games and strobe glasses. The results will allow us to understand which visual training is more beneficial for improving dynamic visual acuity in athletes.

ELIGIBILITY:
Inclusion Criteria:

* No strabismus and/or amblyopia.
* Not presenting accommodative difficulties or difficulties in ocular convergence.

Exclusion Criteria:

* Presence of amblyopia and strabismus, accommodative insufficiency, convergence insufficiency
* Be federated in any sport in which they train more than 3 hours a week in the past and previous year (1 year ago) from the day of the experimental measurements.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Dynamic Visual Acuity | Before the intervention
  Dynamic Visual Acuity 1.0 m/s and contrast 100%
Dynamic Visual Acuity | Immediately after the intervention
  Dynamic Visual Acuity 1.0 m/s and contrast 100%
Dynamic Visual Acuity | 1 month
  Dynamic Visual Acuity 1.0 m/s and contrast 100%
Dynamic Visual Acuity | Before the intervention
  Dynamic Visual Acuity 1.0 m/s and contrast 10%
Dynamic Visual Acuity | Immediately after the intervention
  Dynamic Visual Acuity 1.0 m/s and contrast 10%
Dynamic Visual Acuity | 1 month
  Dynamic Visual Acuity 1.0 m/s and contrast 10%
Dynamic Visual Acuity | Before the intervention
  Dynamic Visual Acuity 0,5 m/s and contrast 100%
Dynamic Visual Acuity | Immediately after the intervention
  Dynamic Visual Acuity 0,5 m/s and contrast 100%
Dynamic Visual Acuity | 1 month
  Dynamic Visual Acuity 0,5 m/s and contrast 100%
Dynamic Visual Acuity | Before the intervention
  Dynamic Visual Acuity 0,5 m/s and contrast 10%
Dynamic Visual Acuity | Immediately after the intervention
  Dynamic Visual Acuity 0,5 m/s and contrast 10%
Dynamic Visual Acuity | 1 month
  Dynamic Visual Acuity 0,5 m/s and contrast 10%

SECONDARY OUTCOMES:
Posner task | Before the intervention
  Change of attention
Posner task | Immediately after the intervention
  Change of attention
Posner task | 1 month
  Change of attention
Go - No - Go task | Before the intervention
  Selective attention and response control
Go - No - Go task | Immediately after the intervention
  Selective attention and response control
Go - No - Go task | 1 month
  Selective attention and response control
Multiple object tracking (MOT) | Before the intervention
  Simultaneously monitor multiple moving objects.
Multiple object tracking (MOT) | Immediately after the intervention
  Simultaneously monitor multiple moving objects.
Multiple object tracking (MOT) | 1 month
  Simultaneously monitor multiple moving objects.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green CS, Bavelier D. Action-video-game experience alters the spatial resolution of vision. Psychol Sci. 2007 Jan;18(1):88-94. doi: 10.1111/j.1467-9280.2007.01853.x. PMID 17362383
- [Background] Feng J, Spence I. Playing action video games boosts visual attention. In: Video game influences on aggression, cognition, and attention. Springer; 2018. p. 93-104
- [Background] Green CS, Bavelier D. Learning, attentional control, and action video games. Curr Biol. 2012 Mar 20;22(6):R197-206. doi: 10.1016/j.cub.2012.02.012. PMID 22440805
- [Background] Green CS, Bavelier D. Action video game training for cognitive enhancement. Curr Opin Behav Sci. 2015;4:103-8.
- [Background] Green CS, Li R, Bavelier D. Perceptual learning during action video game playing. Top Cogn Sci. 2010 Apr;2(2):202-16. doi: 10.1111/j.1756-8765.2009.01054.x. Epub 2009 Oct 30. PMID 25163784
- [Background] Li L, Chen R, Chen J. Playing Action Video Games Improves Visuomotor Control. Psychol Sci. 2016 Aug;27(8):1092-108. doi: 10.1177/0956797616650300. Epub 2016 Jul 8. PMID 27485132
- [Background] Green CS, Bavelier D. Action video game modifies visual selective attention. Nature. 2003 May 29;423(6939):534-7. doi: 10.1038/nature01647. PMID 12774121
- [Background] Dye MW, Green CS, Bavelier D. Increasing Speed of Processing With Action Video Games. Curr Dir Psychol Sci. 2009;18(6):321-326. doi: 10.1111/j.1467-8721.2009.01660.x. PMID 20485453
- [Background] Wilkins L, Appelbaum LG. An early review of stroboscopic visual training: insights, challenges and accomplishments to guide future studies. Int Rev Sport Exerc Psychol. 2020;13(1):65-80.
- [Background] Clark JF, Ellis JK, Bench J, Khoury J, Graman P. High-performance vision training improves batting statistics for University of Cincinnati baseball players. PLoS One. 2012;7(1):e29109. doi: 10.1371/journal.pone.0029109. Epub 2012 Jan 19. PMID 22276103
- [Background] Wilkins L, Nelson C, Tweddle S. Stroboscopic visual training: A pilot study with three elite youth football goalkeepers. Journal of Cognitive Enhancement. 2018;2:3-11.
- [Background] Holliday J. Effect of stroboscopic vision training on dynamic visual acuity scores: Nike Vapor Strobe® Eyewear. 2013
- [Background] Wilkins L, Gray R. EFFECTS OF STROBOSCOPIC VISUAL TRAINING ON VISUAL ATTENTION, MOTION PERCEPTION, AND CATCHING PERFORMANCE. Percept Mot Skills. 2015 Aug;121(1):57-79. doi: 10.2466/22.25.PMS.121c11x0. Epub 2015 Jun 30. PMID 26126135